CLINICAL TRIAL: NCT04781387
Title: A Phase 2, Randomized, Double-Blind, Comparator-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of CRS3123 Compared With Oral Vancomycin in Adults With Clostridioides Difficile Infection
Brief Title: Evaluation of CRS3123 vs. Oral Vancomycin in Adult Patients With Clostridioides Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crestone, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-0021; 75N93019C00056 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2021-01-19; First posted 2021-03-04 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Clostridioides Difficile Infection
Keywords: CDI; Cdiff Infection; Clostridiodes difficile infection; Cdiff
MeSH Terms: conditions — Clostridium Infections | interventions — REP 3123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CRS3123 200 milligram (Experimental): CRS3123 200 milligram dose (400 mg/day) given orally at approximately 6-hour intervals for 10 days.
  Due to the difference in dosing schedules between CRS3123 (twice a day) and the standard of care vancomycin (four times a day) and appearance of study drugs used in the 3 Arms, placebo will be used to match the total number of capsules in each arm.
  Interventions: Drug: CRS3123
- CRS3123 400 milligram (Experimental): CRS3123 400 milligram dose (800 mg/day) given orally at approximately 6-hour intervals for 10 days.
  Due to the difference in dosing schedules between CRS3123 (twice a day) and the standard of care vancomycin (four times a day) and appearance of study drugs used in the 3 Arms, placebo will be used to match the total number of capsules in each arm.
  Interventions: Drug: CRS3123
- Vancomycin 125 milligram (Active Comparator): Vancomycin 125 milligram dose (500 mg/day) given orally at approximately 6-hour intervals for 10 days.
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: CRS3123 — Study drug dosed PO BID for a total of 10 days
  Arms: CRS3123 200 milligram; CRS3123 400 milligram
Drug: Active Comparator — Active comparator dosed PO QID for 10 days
  Arms: Vancomycin 125 milligram

SUMMARY:
The purpose of this research is to evaluate the primary objectives of safety and efficacy (rate of clinical cure) of 2 dosages of CRS3123 (200 mg and 400 mg) administered orally (po) twice daily (bid) and vancomycin administered 125 mg PO 4 times daily (qid) in adults > or equal to 18 years of age with a primary episode or first recurrence of CDI. The study will investigate the plasma concentrations and HRQoL outcomes of CRS3123 and additional efficacy endpoints as secondary objectives.

ELIGIBILITY:
Inclusion Criteria

1. Adults, ≥ 18 years of age.
2. More than or equal to 3 diarrheal (Bristol Stool Scale scores 5, 6, or 7) stools/day in a 24-hour period during screening prior to randomization and in the judgment of the investigator that C. difficile is the likely causative agent for the diarrhea.
3. Stool positive for C. difficile Toxin A and/or B antigen using an FDA or Health Canada approved/cleared EIA or ELISA laboratory test.
4. Participants with a primary episode or first recurrence of CDI are eligible.
5. In the judgment of the investigator, the expectation that the participant will survive with effective antibiotic therapy and appropriate supportive care for the anticipated duration of the study.
6. Female participants of childbearing potential must not be pregnant, plan to become pregnant during the study, or be breastfeeding; and must be willing to commit to either sexual abstinence or use highly effective methods of birth control contraception from screening through Day 70.
7. Males must use a condom and spermicide from screening through Day 70 (if the female partner(s) is of childbearing potential) and must not donate sperm from screening through Day 70.
8. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria

1. Participants with any of the following conditions:

   1. Intractable vomiting preventing oral medication intake
   2. Severe underlying disease with an expected survival time less than the duration of the study (approximately 70 days).
   3. More than 1 prior CDI occurrence within the last 3 months or more than 2 prior episodes of CDI in the last 12 months.
   4. A history of a recent CDI episode within 3 months prior to enrollment that was non- responsive to vancomycin.
   5. In the investigator's opinion, the participant is anticipated to require oral or intravenous systemic antibiotic therapy for a non-CDI infection between screening and Day 70.
   6. Inflammatory bowel disease (Crohn's disease or ulcerative colitis), uncorrected Hirschsprung's disease, short gut syndrome, or any other condition known to significantly impact bowel motility and/or malabsorption.
   7. Any other known pathogen associated with diarrhea.
   8. Life-threatening or fulminant CDI as defined by IDSA/SHEA Guidelines.
   9. Colonic perforation.
   10. Need for concurrent laxatives or tube feeds, toxin binders, bile acid sequestrants during the study. Microbiota restoration therapy (MRT) or any phage therapy within 1 year of randomization. Receipt of bezlotoxumab within 3 months of randomization.
   11. Participants treated with another antimicrobial agent directed at the current episode of CDI (metronidazole, fidaxomicin, rifaximin, tigecycline, or oral vancomycin) for >24 hours of treatment within the 3 days prior to randomization will not be eligible for enrollment.
2. Pregnant or breastfeeding women.
3. Receipt of any investigational medication during the last month (30 days or 5 half lives, whichever is longer) prior to randomization.
4. Active and uncontrolled HIV with CD4 <200/mm3.
5. Presence of active malignancy undergoing chemotherapy that is expected to cause significant immunosuppression, hematologic malignancy undergoing induction chemotherapy, or recent bone marrow or solid organ transplant (within 1 month prior to randomization) undergoing treatment with medications for the rejection of transplantation. In the investigator's opinion, is expected not to survive through the duration of the study (approximately 70 days) due to complications of the malignancy, or in the investigator's opinion will require oral or intravenous systemic antibiotic therapy during the study for malignancy related conditions.
6. Severe neutropenia defined as ANC <500 cells/mm3
7. Severe hepatic impairment at screening including clinical signs of cirrhosis, end-stage hepatic disease (eg, ascites, hepatic encephalopathy), or Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3x upper limit of normal (ULN) or total bilirubin ≥ 2x ULN.
8. Any other surgical or medical condition (including a clinically significant laboratory abnormality) as determined by the investigator or the medical monitor, that could interfere with the participant's ability to participate in the study, the administration of study treatment, and/or the interpretation of study results that, in the investigator's opinion, may confound study assessments or study procedures.
9. Known hypersensitivity to CRS3123 or oral vancomycin.
10. An employee of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as a family member of the employee or the investigator.
11. Unwillingness to stop consuming non-dietary probiotics from randomization to Day 70.
12. Participants currently taking digoxin within 1 week of screening.
13. Unwillingness to refrain from consumption of grapefruit and its juices as well as nutraceutical supplements containing curcumin from randomization until 24 hours after EOT.
14. Unwillingness to stop use of anti-diarrheals from randomization to Day 70.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urs Ochsner, PhD, Principal Investigator — Crestone, Inc
Locations (20):
- United States (18):
  - 131, Fullerton, California
  - 117, Lancaster, California
  - 143, Mission Hills, California
  - 138, Orange, California
  - 146, Miami, Florida
  - 122, Miami, Florida
  - 140, Marietta, Georgia
  - 110, Idaho Falls, Idaho
  - 129, Winfield, Illinois
  - 130, Royal Oak, Michigan
  - 139, Weldon Spring, Missouri
  - 128, Butte, Montana
  - 134, The Bronx, New York
  - 147, Chapel Hill, North Carolina
  - 114, Uniontown, Pennsylvania
  - 104, Cedar Park, Texas
  - 123, Houston, Texas
  - 101, San Antonio, Texas
- Canada (2):
  - 116, Calgary, Alberta
  - 120, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louie T, Ribble W, Boccumini L, Johnson K, De Groote MA, Day J, Mason C, Sun X, Freeman J, Gu K, Tillotson G, Wilcox MH, Janjic N, Jarvis TC, Nayak SU, Ochsner UA, Bruss JB. Safety and efficacy of CRS3123 in adults with a primary episode or first recurrence of Clostridioides difficile infection: a phase 2, randomised, double-blind, multicentre, vancomycin-controlled study. Lancet Infect Dis. 2026 Jan 22:S1473-3099(25)00721-2. doi: 10.1016/S1473-3099(25)00721-2. Online ahead of print. PMID 41581516

RESULTS

PARTICIPANT FLOW:
Groups:
- CRS3123 200 Milligram: CRS3123 200 milligram dose (400 mg/day) given orally at approximately 12-hour intervals for 10 days.
- CRS3123 400 Milligram: CRS3123 400 milligram dose (800 mg/day) given orally at approximately 12-hour intervals for 10 days.
Period: Overall Study
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Started | 14 | 15 | 14
Completed | 12 | 15 | 13
Not Completed | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram | Total
Number analyzed (Participants) | 14 | 15 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 7 | 27
  >=65 years | 4 | 5 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 10 | 33
  Male | 2 | 4 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 8 | 13
  Not Hispanic or Latino | 13 | 11 | 6 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 11 | 14 | 13 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 6 | 5 | 15
  United States | 10 | 9 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Cure at the Test of Cure [TOC] Visit in the Intent-to-treat [ITT] Population
Description: Clinical cure is defined as survival through TOC/Day 12 and resolution of diarrhea (i.e., <3 unformed bowel movements [UBM] [Bristol Stool Scale score of 5, 6, or 7] at end-of-treatment (EOT)/Day 10 with maintenance of resolution through TOC/Day 12 and no further requirement for treatment of CDI through TOC/Day 12. Numbers reported below indicate participants from each cohort that were clinical cures, clinical failures, or indeterminate at the TOC/Day 12 visit.
Time Frame: TOC/Day 12
Population: ITT: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 14 | 15 | 14
Participants
  Clinical Cure | 13 | 15 | 13
  Clinical Failure | 0 | 0 | 0
  Indeterminate | 1 | 0 | 1

2. Secondary Outcome: Rate of Clinical Cure at Test of Cure (TOC) in the Microbiological-ITT (mITT) Population
Description: Clinical cure is defined as survival through TOC/Day 12 and resolution of diarrhea (i.e., <3 unformed bowel movements [UBM] [Bristol Stool Scale score of 5, 6, or 7] at end-of-treatment (EOT)/Day 10 with maintenance of resolution through TOC/Day 12 and no further requirement for treatment of CDI through TOC/Day 12. Numbers reported below indicate participants from each cohort that were clinical cures, clinical failures, or indeterminate at the TOC/Day12 visit.
Time Frame: TOC/Day 12
Population: mITT: Participants in the ITT population who have Cdiff isolated in culture and who are Cdiff toxin positive from a screening or Day 1 fecal sample
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 13 | 14 | 13
Participants
  Clinical Cure | 12 | 14 | 13
  Clinical Failure | 0 | 0 | 0
  Indeterminant | 1 | 0 | 0

3. Secondary Outcome: Rate of Clinical Cure at Test of Cure (TOC) in the Per Protocol (PP) and Microbiologically Evaluable (ME) Populations
Description: as for outcome 2
Time Frame: TOC/Day 12
Population: PP: Participants who receive at least 80% of the planned doses, receive no concomitant systemic antibiotics, prohibited probiotic or anti-diarrheal medication from randomization through TOC, and have an investigator assessment of clinical response at TOC; ME: Participants in the PP and Micro-ITT populations
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  PP: Clinical Cure | 12 | 14 | 13
  PP: Clinical Failure | 0 | 0 | 0
  PP: Indeterminate | 0 | 0 | 0
  ME: Clinical Cure | 12 | 14 | 13
  ME: Clinical Failure | 0 | 0 | 0
  ME: Indeterminate | 0 | 0 | 0

4. Secondary Outcome: Rate of Total Relief of Symptoms of Clostridioides Difficile Infection at Test of Cure (TOC) in the Microbiological-ITT (mITT) Population
Description: Total relief of symptoms at TOC/Day 12 is defined as resolution (< 3 per day) of unformed bowel movements, an investigator's assessment of clinical cure, and the resolution of signs or symptoms of CDI recorded at baseline. Numbers reported below indicate participants from each cohort that had total relief of symptoms at TOC/Day 12 and those that did not.
Time Frame: TOC/Day 12
Population: mITT: Participants in the ITT population who have Cdiff isolated in culture and are Cdiff toxin positive from a screening or Day 1 fecal sample
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 13 | 14 | 13
Participants
  Total Relief of Symptoms -- Yes | 11 | 14 | 12
  Total Relief of Symptoms -- No | 1 | 0 | 1
  Total Relief of Symptoms -- Indeterminate | 1 | 0 | 0

5. Secondary Outcome: Rate of Total Relief of Symptoms of Clostridioides Difficile Infection at Test of Cure (TOC) in the Per Protocol (PP) and Microbiologically Evaluable (ME) Populations
Description: as for outcome 4
Time Frame: TOC/Day 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  PP: Total Relief of Symptoms -- Yes | 11 | 14 | 12
  PP: Total Relief of Symptoms -- No | 1 | 0 | 1
  PP: Total Relief of Symptoms -- Indeterminate | 0 | 0 | 0
  ME: Total Relief of Symptoms -- Yes | 11 | 14 | 12
  ME: Total Relief of Symptoms -- No | 1 | 0 | 1
  ME: Total Relief of Symptoms -- Indeterminate | 0 | 0 | 0

6. Secondary Outcome: Time to Resolution of Diarrhea Through Test of Cure (TOC) in the Microbiological-ITT (mITT) Population
Description: The time to resolution of diarrhea is defined as the time elapsed from the first dose of study treatment to the last unformed bowel movement before 2 consecutive days of < 3 unformed bowel movements (Bristol Stool Scale score of 5, 6, or 7) per day through TOC/Day 12. Values reported below are median days to resolution for each cohort.
Time Frame: Study Day 1 until the date of documented resolution, assessed up to TOC/Day 12
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 13 | 14 | 13
Days | 2.6 [0.9 to 3.4] | 3.9 [1.2 to 4.6] | 1.9 [0.0 to 4.7]

7. Secondary Outcome: Time to Resolution of Diarrhea Through Test of Cure (TOC) in the Per Protocol (PP) and Microbiologically Evaluable (ME) Populations
Description: as for outcome 6
Time Frame: Study Day 1 until the date of documented resolution, assessed up to TOC/Day 12
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Days
  PP | 2.7 [0.9 to 4.0] | 3.9 [1.2 to 4.6] | 1.9 [0.0 to 4.7]
  ME | 2.7 [0.9 to 4.0] | 3.9 [1.2 to 4.6] | 1.9 [0.0 to 4.7]

8. Secondary Outcome: Rate of Early Recurrence of Clostridioides Difficile Infection Through Day 40 in the Microbiological-ITT (mITT) Population
Description: Rate of early recurrence of C. difficile infection (CDI) is defined as a new episode of diarrhea (≥ 3 unformed bowel movements [Bristol Stool Scale score of 5, 6, or 7] in a 24-hour period) with a positive toxin result and requires retreatment for CDI before Day 40. The table below shows the number of participants per cohort that experienced a recurrence before Day 40 and those that did not. Only participants that were clinical cures at TOC/Day 12 were included in the analysis.
Time Frame: Post TOC/Day 12 visit through Day 40
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  Recurrence -- Yes | 0 | 1 | 3
  Recurrence -- No | 12 | 13 | 10

9. Secondary Outcome: Rate of Early Recurrence of Clostridioides Difficile Infection Through Day 40 in the Microbiologically Evaluable (ME) Population
Description: as for outcome 8
Time Frame: Post TOC/Day 12 visit through Day 40
Population: ME: Participants in the PP and Micro-ITT populations
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  Recurrence -- Yes | 0 | 1 | 3
  Recurrence -- No | 12 | 13 | 10

10. Secondary Outcome: Rate of Late Recurrence of Clostridioides Difficile Infection (Between Day 40 and Day 70) in the Microbiological-ITT (mITT) Population
Description: Rate of late recurrence of CDI is defined as a new episode of diarrhea (≥ 3 unformed bowel movements [Bristol Stool Scale score of 5, 6, or 7] in a 24-hour period), with a positive toxin result and requires retreatment of CDI between Day 40 and Day 70. The table below shows the number of participants per cohort that experienced a recurrence between Day 40 and Day 70 and those that did not. Analysis populations for this assessment only includes participants that had an investigator assessment of clinical cure at TOC/Day 12. Participants that were indeterminate at TOC/Day 12 or recurrent prior to Day 40 were excluded.
Time Frame: Day 40 - Day 70
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 13 | 10
Participants
  Recurrence -- Yes | 0 | 1 | 0
  Recurrence -- No | 12 | 12 | 10

11. Secondary Outcome: Rate of Late Recurrence of Clostridioides Difficile Infection (Between Day 40 and Day 70) in the Microbiologically Evaluable (ME) Population
Description: as for outcome 10
Time Frame: Day 40 - Day 70
Population: ME: Participants in the PP and Micro-ITT populations
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 13 | 10
Participants
  Recurrence -- Yes | 0 | 1 | 0
  Recurrence -- No | 12 | 12 | 10

12. Secondary Outcome: Rate of Recurrence of Clostridioides Difficile Infection Through Day 70 in the Microbiological-ITT (mITT) Population
Description: Rate of recurrence of CDI is defined as a new episode of diarrhea (≥3 unformed bowel movements [Bristol Stool Scale score of 5, 6, or 7] in a 24-hour period) with a positive toxin result and requires retreatment for CDI at any point between TOC/Day 12 and Day 70. The table below shows the number of participants per cohort that experienced a recurrence between TOC/Day 12 and Day 70 and those that did not. Analysis populations for this assessment only includes participants that had an investigator assessment of clinical cure at TOC/Day 12.
Time Frame: Post TOC/Day 12 visit through Day 70
Population: Micro-ITT: All participants in the ITT population who have C. difficile isolated in culture and who are C. difficile toxin positive at the central laboratory from a screening or Day 1 fecal sample
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  Recurrence -- Yes | 0 | 2 | 3
  Recurrence -- No | 12 | 12 | 10

13. Secondary Outcome: Rate of Recurrence of Clostridioides Difficile Infection Through Day 70 in the Microbiologic Evaluable (ME) Population
Description: as for outcome 12
Time Frame: Post TOC/Day 12 visit through Day 70
Population: ME: Participants in the PP and Micro-ITT populations.
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  Recurrence -- Yes | 0 | 2 | 3
  Recurrence -- No | 12 | 12 | 10

14. Secondary Outcome: Rate of Global Cure in the Microbiological-ITT (mITT) Population
Description: Global cure is defined as a clinical cure at TOC/Day 12 without recurrence through Day 40. The table below shows the number of participants per cohort that experienced a recurrence between TOC/Day 12 and Day 40 and those that did not.
Time Frame: Post TOC/Day 12 visit through Day 40
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 13 | 14 | 13
Participants
  Global cure -- Yes | 12 | 13 | 10
  Global Cure --No | 1 | 1 | 3

15. Secondary Outcome: Rate of Global Cure in the Per Protocol (PP) and Microbiologically Evaluable (ME) Populations
Description: as for outcome 14
Time Frame: Post TOC/Day 12 visit through Day 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
Number analyzed (Participants) | 12 | 14 | 13
Participants
  PP: Global Cure -- Yes | 12 | 13 | 10
  PP: Global Cure -- No | 0 | 1 | 3
  ME: Global Cure -- Yes | 12 | 13 | 10
  ME: Global Cure -- No | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: Safety assessments were performed at each visit from screening/Day -1 to the final follow-up visit on Day 70
Description: Adverse event information is reported by number and frequency per cohort by: 1) All-Cause Mortality: All anticipated and unanticipated deaths due to any cause, 2) Serious Adverse Events: All anticipated and unanticipated serious adverse events, grouped by organ system, and 3) Other Adverse Events: Anticipated and unanticipated events (not included in the serious adverse event table) that exceed a frequency threshold of 4% within any arm of the clinical study, grouped by organ system
Arm/Group | CRS3123 200 Milligram | CRS3123 400 Milligram | Vancomycin 125 Milligram
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 8/14 | 7/15 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRS3123 200 Milligram (N=14) | CRS3123 400 Milligram (N=15) | Vancomycin 125 Milligram (N=14)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRS3123 200 Milligram (N=14) | CRS3123 400 Milligram (N=15) | Vancomycin 125 Milligram (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or other public disclosure, written or oral, relating to or derived from the Confidential Information, or relating to the Consultant's work with Crestone, shall be provided by the Consultant to Crestone at least 90 days prior to submission for publication or other disclosure. Crestone shall review the publication or other disclosure within a reasonable period of time and inform the Consultant as to whether or not Crestone consents to publication or other disclosure.

DOCUMENTS (3):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04781387/Prot_001.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT04781387/SAP_002.pdf
  • Informed Consent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT04781387/ICF_004.pdf